CLINICAL TRIAL: NCT07366463
Title: Integrating Hepatological, Nutritional, and Cognitive Behavioral Therapy-based Psychological Support is an Effective Multidisciplinary Approach to Improve Long-term Clinical Outcomes in the Management of MASLD Patients: a Randomized Clinical Trial [The "CoCoNut" Study]
Brief Title: Integrating Hepatological, Nutritional, and Psychological Support as a Multidisciplinary Management to Improve Long-term Clinical Outcomes in MASLD
Acronym: CoCoNut
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Alessandro Federico, Full Professor, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0016368/i
Record Dates: First submitted 2025-12-30; First posted 2026-01-26 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: MASLD - Metabolic Dysfunction-Associated Steatotic Liver Disease; MASLD; Cardiovascular Events
Keywords: Multidisciplinary; Nutrition; Cognitive behavioral therapy; Personalized medicine
MeSH Terms: interventions — Nutritional Support; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: In this randomized controlled trial (RCT), patients admitted to the Hepatogastroenterology Unit of the "Luigi Vanvitelli" University Hospital presenting with a diagnosis of MASLD will consecutively enrolled and randomized to receive hepatologist counseling with generic lifestyle recommendations (Group A - "Hep"), hepatologist counseling with the integration of tailored lifestyle recommendations, including personalized physical exercise and dietary plan, provided by a nutritionist (Group B - "Hep + Nut"), or hepatologist counseling with the integration of tailored lifestyle recommendations, including personalized physical exercise and dietary plan, provided by a nutritionist, combined with CBT program-based psychological support, offered by a psychologist specialist, for a period of 18 months (Group C - "Hep + Nut + Psy"). .
  Groups A and B constituted the standard of care, while Group C, receiving the multidisciplinary triple approach ("Co-Co-Nut" ), represented the experimental.
Who Masked: Care Provider, Investigator
Masking Description: To conceal the allocation of the patients, block sizes will not be disclosed to investigators enrolling patients, and investigators recruiting patients will not know to which group the next patient will be assigned. For this purpose, investigators not involved in patient enrollment (i.e., external investigators) will prepare a sequence of numbered, opaque, sealed envelopes containing the patient's group. To prevent tampering, the list will remain inaccessible, and the envelopes will be opened sequentially after enrolling the patient and obtaining consent.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A - "Hep" (Active Comparator): Hepatologist counseling providing generic lifestyle recommendations
  Interventions: Behavioral: Hepatologic-provided recommendations
- Group B - "Hep + Nut" (Active Comparator): Hepatologist counseling with the integration of tailored lifestyle recommendations, including personalized physical exercise and dietary plan, provided by a nutritionist
  Interventions: Behavioral: Hepatologic-provided recommendations; Behavioral: Nutritional support
- Group C - "Hep + Nut + Psy" (Experimental): Hepatologist counseling with the integration of tailored lifestyle recommendations, including personalized physical exercise and dietary plan, provided by a nutritionist, combined with cognitive behavioral therapy (CBT) program-based psychological support, offered by a psychologist specialist
  Interventions: Behavioral: Hepatologic-provided recommendations; Behavioral: Nutritional support; Behavioral: Psychological support

INTERVENTIONS:
Behavioral: Hepatologic-provided recommendations — Hepatologic counseling will be offered every six months to individuals belonging to all study groups. These specialists-provided check-ups consisted of recording, at baseline, demographics and, at baseline and every six months, collecting anthropometrical, biochemical, clinical (including the assessment of previous cardiovascular events and the determination of individual cardiovascular risk), and body composition data, as well as evaluating the liver disease progression by using Noninvasive tools (NITs) (Fibroscan CAP).
  Moreover, at baseline, the hepatologist, after assessing the initial compliance of each individual with the Mediterranean diet and active physical exercise, by respectively adopting the MDS questionnaire and the IPAQ-SF score questionnaire, also recommended, for the entire duration of the study, generic lifestyle changes, including a Mediterranean diet style, and proper physical activity (> 150 min/week of moderate - or 75 min/week of vigorous physical activity).
Behavioral: Nutritional support — Nutritional counseling by a specialist will be provided on a semestral basis, scheduled on the same day as the hepatology follow-up visits, although conducted separately and after the hepatology consultation, and was offered exclusively to patients in Groups B and C. In these occasions, specialised anamnesis will be performed (including the investigation of general dietary habits, food allergies, and taste preferences), as well as the multicompartmental BIA-assessed body composition results will be properly interpreted to design, and eventually dynamically change along the duration of the study, a personalised dietary plan with a tailored physical activity strategy (integrating the generic recommendations received by the hepatologists), as well as to establish, and periodically revaluate, individual body composition outcomes.
  Arms: Group B - "Hep + Nut"; Group C - "Hep + Nut + Psy"
Behavioral: Psychological support — The psychological intervention will be structured in sequential phases to enhance disease awareness, coping skills, and adherence to lifestyle changes. The first 90-minute session will include a comprehensive personal, familial, and physiological assessment, with systematic evaluation of social determinants of health using a dedicated CRF. The psychologist will assess disease awareness, quality of life, motivation for change, and treatment expectations. Emotional and cognitive components will be explored through interviews and standardized tools (BAI, BDI-II). Individualized therapeutic goals will be jointly defined. Weekly 60-minute sessions over six months will address previous behavioural change attempts, barriers, facilitators, and strategy refinement. Motivation will be continuously monitored according to the Transtheoretical Model. Semiannual follow-up sessions will reassess progress and address emotional or situational challenges.
  Other Names: Cognitive behavioral therapy
  Arms: Group C - "Hep + Nut + Psy"

SUMMARY:
Metabolic dysfunction associated Steatotic Liver Disease (MASLD) is frequently complicated by cardiometabolic (CMR) comorbidities, and prognosis is substantially influenced by acute cardiovascular events (ACE). Although several pharmacological approaches target CMR risk factors, lifestyle modification remains the cornerstone of management. However, adherence to dietary behavioral prescriptions is often poor, and the influence of sociodemographic determinants on compliance remains unclear. Moreover, the long-term real-life impact of behavioral and motivational support in MASLD is insufficiently characterized.

This randomized controlled trial aims to evaluate the effectiveness of a multidisciplinary management (including Hepatological counseling, Nutrition intervention, and Psychological support) in improving clinical MASLD outcomes, by increasing adherence to specialist-tailored recommendations.

DETAILED DESCRIPTION:
Metabolic dysfunction-associated Steatotic Liver disease (MASLD) represents a predominant hepatopathy worldwide, as well as a complex systemic condition complicated by various extra-hepatic dysmetabolic manifestations.

Among these, acute cardiovascular events represent a serious burden, drastically increasing mortality rates, emphasizing the absolute need for holistic and multidisciplinary treatment strategies.

Even though several pharmacological approaches have been proposed, targeting the different dysmetabolic manifestations, lifestyle changes remain the paramount intervention for patients with simple steatosis. However, adherence to dietary and behavioral recommendations is often poor. Growing evidence highlights the importance of cognitive behavioral therapy (CBT) in supporting these recommendations. However, the real benefits of providing motivational support to individuals with MASLD remain largely unexplored in real-world applications.

This randomized controlled trial aims to evaluate the effectiveness of a multidisciplinary approach (integrating Hepatological counseling, Nutrition intervention, and Psychological support) in improving long-term clinical MASLD outcomes, by increasing adherence to specialist-tailored recommendations, as well as to investigate the social determinants impacting on the loss of compliance with this strategy.

MASLD patients will be consecutively enrolled and randomized into three Groups:

* Group A - following generic hepatologist-provided advice ("H"),
* Group B- also receiving a nutritionist-prescribed individualized intervention ("HN")
* Group C- receiving an approach which additionally involves cognitive/behavioral-based psychological support ("HNP")

Groups A and B represent the "standard of care" cohort, while Group B represents the "experimental" cohort.

Baseline anthropometric, biochemical, clinical, liver stiffness (LSM), controlled attenuation parameter (CAP), lifestyle habits (including dietary and physical exercise), and body composition values will be recorded.

Along 18 months:

* Semestral hepatological (for all), nutritional (H and HN), and psychological (HNP) follow-ups reassess variables and evaluated compliance.
* Acute Cardiovascular events will be recorded

ELIGIBILITY:
Inclusion Criteria:

* age between 40 and 79 years,
* a diagnosis of MASLD, configured by the presence of hepatic steatosis (proven by instrumental and/or histological methods), with at least one of the five cardiometabolic risk factors (CMRFs) as established by the updated multi-society Delphi consensus proposed criteria,
* willingness to sign a valid informed consent

Exclusion Criteria:

* unavailability or inability to express written consent,
* chronic liver diseases other than MASLD/overlap ongoing causes (including chronic hepatitis B virus infection, chronic hepatitis C virus infection, autoimmune hepatitis, chronic cholestasis, genetic diseases determining steatosis, and alcohol-related liver disorder assumed in the evidence of a history of alcohol intake greater than 20 g/day or 140 g/week),
* administration of liver-damaging (Drug-induced liver Injury) (DILI) / hepatic steatosis inducing drugs (Drug-Induced Fatty Liver Disease) (DIFLD),
* hepatoprotective drugs administration,
* consumption of hypoglycemic, hypolipidemic, and weight loss agents, as well as any drug known to influence liver function,
* neoplasms,
* chronic systemic inflammatory diseases,
* eating disorders (ED)
* other psychiatric disorders potentially invalidating the consent.

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-20 (Actual)

PRIMARY OUTCOMES:
Body Weight reduction | From enrollment to the end of intervention at 18 months
  The primary endpoint of this study was to highlight a significantly higher proportion (at least > 15%) of patients obtaining (intermediate time-point, i.e., after 12 months), and maintaining (end of the study, i.e., after 18 months), a reduction of at least 10% in body weight in the experimental cohort compared with the standard of care

SECONDARY OUTCOMES:
Variations in anthropometric parameters | From enrollment to the end of intervention at 18 months
  After 18 months, at the end of the study, in the experimental cohort compared with the standard of care, to report a statistically significant improvement of Body Mass Index (BMI) and Waist-to-hip ratio (WHR)].
Different risk of acute cardiovascular events | From enrollment to the end of intervention at 18 months
  In the experimental cohort compared with the standard of care, to highlight significant changes in cardiovascular risk by using the Atherosclerotic Cardiovascular Disease (ASCVD) risk score, adopting the calculator available online on the American College of Cardiology website (https://tools.acc.org/ascvd-risk-estimator-plus) (accessed on 4th June 2024), considering > 7.5% the threshold defining a significant risk.
Variations in metabolic variables (glycometabolic) | From enrollment to the end of intervention at 18 months
  After the 18 months, at the end of the study, in the experimental cohort compared with the standard of care, to report a statistically significant improvement of Homeostatic Model Assessment for Insulin Resistance (HOMA-IR),
Variations in metabolic parameters (lipidic variables) | From enrollment to the end of intervention at 18 months
  After the 18 months, at the end of the study, in the experimental cohort compared with the standard of care, to report a statistically significant improvement of high-density lipoprotein cholesterol (HDL)],
Variations in body composition | From enrollment to the end of intervention at 18 months
  After 18 months, at the end of the study, in the experimental cohort compared with the standard of care, to report a statistically significant improvement of body composition parameters [free-fat mass (FFM) and fat mass (FM)].
Variations in Liver Stiffness | From enrollment to the end of intervention at 18 months
  After the 18 months, at the end of the study, in the experimental cohort compared with the standard of care, to report a statistically significant improvement of Liver Stiffness Measurement (LSM).
Variations in Controlled Attenuation Parameter (CAP) | From enrollment to the end of intervention at 18 months
  After the 18 months, at the end of the study, in the experimental cohort compared with the standard of care, to report a statistically significant improvement of Controlled Attenuation Parameter (CAP).

OTHER OUTCOMES:
Relationship between anxiety severity and levels of compliance with the intervention | From enrollment to the end of intervention at 18 months
  To reveal a significant correlation between anxiety levels [Beck Anxiety Inventory (BAI) questionnaire] and levels of compliance with the assigned intervention.
  Note: Adherence to the assigned behavioral intervention is assessed using a 4-item questionnaire specifically developed for this study. The tool is conceptually informed by general adherence principles but is independently created, with original items and scoring, and does not reproduce or rely on the proprietary MMAS-4.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Campania Luigi Vanvitelli, Naples, Campania, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Romeo M, Dallio M, Cipullo M, Coppola A, Mazzarella C, Mammone S, Iadanza G, Napolitano C, Vaia P, Ventriglia L, Federico A. Nutritional and Psychological Support as a Multidisciplinary Coordinated Approach in the Management of Chronic Liver Disease: A Scoping Review. Nutr Rev. 2025 Jul 1;83(7):1327-1343. doi: 10.1093/nutrit/nuaf001. PMID 39992295
- [Result] M. Romeo, M. Dallio, F. Di Nardo, A. Coppola, P. Vaia, C. Napolitano, G. Martinelli, S. Olivieri, M. Niosi, A. Federico, Multidisciplinary management combining hepatologist counseling, cognitive/behavioral therapy, and nutritional support significantly improves clinical outcomes of Metabolic dysfunction-associated Steatotic Liver Disease (MASLD) patients, Digestive and Liver Disease, Volume 56, Supplement 3, 2024, Pages S318-S319, ISSN 1590-8658, https://doi.org/10.1016/j.dld.2024.08.009. (https://www.sciencedirect.com/science/article/pii/S1590865824009289)

DOCUMENTS (1):
  • Informed Consent Form (2023-05-31): https://cdn.clinicaltrials.gov/large-docs/63/NCT07366463/ICF_000.pdf